CLINICAL TRIAL: NCT04777071
Title: 68Ga-PSMA-11 PET in Patients With Prostate Cancer
Brief Title: An Investigational Scan (68Ga-PSMA-11 PET) for the Imaging of Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RG1007462; NCI-2020-02612 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10512 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Castration-Resistant Prostate Carcinoma; Prostate Adenocarcinoma; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
Keywords: Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/CT, PET/MR) (Experimental): Patients receive gallium Ga 68-labeled PSMA-11 IV over 60-75 minutes then undergo PET/CT or PET/MR scan over 2-4 minutes per bed position at baseline. Patients receiving systemic therapy undergo an additional 68Ga-PSMA-11 PET/CT or PET/MR scan 12 weeks after initiating therapy. Patients may also undergo CT and bone scan during screening and on study.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Bone Scan; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Magnetic Resonance Imaging — Undergo PET/MR scan
  Other Names: MRI; MR Imaging; NMRI; nuclear magnetic resonance imaging
Procedure: Bone Scan — Undergo bone scan
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This trial studies how well 68Ga-PSMA-11 PET scan works in imaging patients with prostate cancer. Diagnostic procedures, such as 68Ga-PSMA-11 PET may find and diagnose prostate cancer and improve monitoring of treatment response.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive gallium Ga 68-labeled PSMA-11 intravenously (IV) over 60-75 minutes then undergo PET/CT or PET/magnetic resonance (MR) scan over 2-4 minutes per bed position at baseline. Patients receiving systemic therapy undergo an additional 68Ga-PSMA-11 PET/CT or PET/MR scan 12 weeks after initiating therapy. Patients may also undergo CT and bone scan during screening and on study.

After the completion of study, patients are followed up at 60 days, 6 months, and annually up to 5 years or until time of first progression.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven prostate adenocarcinoma
* For the initial staging arm (initial staging cohort), high risk characteristics, including any of the following:

  * Grade group 4-5 and/or
  * PSA > 20 ng/mL
* For patients with biochemical recurrence (biochemical recurrence cohort):

  * Rising PSA after definitive therapy with prostatectomy or targeted local therapy (including but not limited to external beam radiation therapy, brachytherapy, high-frequency ultrasound, and cryotherapy)
  * If post-radical prostatectomy, PSA > 0.2 ng/mL measured > 6 weeks post-operatively and confirmatory persistent PSA greater than 0.2 ng/mL (American Urological Association (AUA) definition for biochemical recurrence
  * If post-radiation therapy, PSA that is equal to, or greater than, a 2 mg/mL rise above PSA nadir (American Society of Radiation Oncology (ASTRO) definition for biochemical recurrence)
* For patients undergoing systemic therapy (treatment monitoring cohort):

  * Diagnosis of metastatic castration-resistant prostate cancer
  * At least one or more measurable ( > 1 cm diameter in short axis) or evaluable lesions by any modality obtained within the past 60 days
  * Planned for treatment with standard of care androgen receptor pathway inhibitor or chemotherapy
* This can include patients who have already undergone a standard of care Ga-68 PSMA PET/CT or PET/MR for determining eligibility for Lu-177 PSMA therapy, for whom the PET/CT or PET/MR did not confirm eligibility for treatment with Lu-177 PSMA, and who are planned to start treatment on chemotherapy or androgen receptor signaling inhibitor (ARSI) within 30 days of the Ga-68 PSMA PET. This can also include patients who have obtained a standard of care Ga-68 PSMA PET/CT or PET/MR for rising PSA to help with restaging prior to starting new treatment with ARSI or chemotherapy, even if Lu-177 PSMA is not being considered at that time. Scan 1 must be completed within 30 days of enrollment. Any patient with an equivocal lesion by conventional imaging, regardless of where they are in the course of evaluation or treatment (equivocal lesion cohort)
* No other malignancy within the past 2 years (with the exception of skin basal cell or cutaneous superficial squamous cell carcinoma, superficial bladder cancer, carcinoma in situ in any location, or Rai Stage 0 chronic lymphocytic leukemia, which are allowed)
* Eastern Cooperative Oncology Group/World Health Organization (ECOG/WHO) performance status grades 0, 1, or 2
* Ability to understand and willingness to provide informed consent

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2030-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in planned management strategy | Baseline up to 1.5 years after the last scan
  Assessed using conventional imaging with executed management strategy incorporating information from first (scan 1) 68Ga-prostate-specific membrane antigen (PSMA)-11 positron emission tomography (PET)/computed tomography (CT), regardless of treatment modality. Will be expressed as the percentage of total patients imaged in which change in management occurred, regardless of treatment modality. The rate of change in management will also be estimated within each group (initial staging, biochemical recurrence, and equivocal lesion cohorts). 95% confidence intervals (CIs) will be used to express precision of the estimates.

SECONDARY OUTCOMES:
Major change in management | Baseline up to 5 years post-scan
  Defined as a change in treatment modality (e.g. change from systemic therapy to radiation therapy). Will compare by planned management strategy using conventional imaging and executed management strategy incorporating information from scan 1 68Ga-PSMA-11 PET/CT, regardless of treatment modality. 95% CIs will be used to express precision of the estimates. This analysis applies to the subjects enrolled in the initial staging (N=30), biochemical recurrence (N=30), and equivocal lesions cohorts (N=43).
Minor change in management | Baseline up to 5 years post-scan
  Defined as changes within a treatment modality (e.g. change in planned radiation field or change in systemic therapy regimen to be used for a patient already planned to receive systemic therapy). Defined as a post-scan change within a treatment modality (e.g. alteration to salvage radiation field). 95% CIs will be used to express precision of the estimates.
68Ga-PSMA-11 standardized uptake value maximum (SUVmax) | Up to 6 weeks after systemic therapy initiation
  Changes in uptake will be compared among all groups using analysis of variance (ANOVA) or the Kruskal-Wallis test and between pairs of groups using the t-test or Wilcoxon rank-sum test.
68Ga-PSMA-11 standard uptake value normalized to lean body mass (SULpeak) | Up to 6 weeks after systemic therapy initiation
  Changes in uptake will be compared among all groups using ANOVA or the Kruskal-Wallis test and between pairs of groups using the t-test or Wilcoxon rank-sum test.
Change in 68Ga-PSMA-11 SUVmax | Baseline up to 6 weeks after systemic therapy initiation
  Expressed as percent (%) change from scan 1. Will be determined and correlated with change in prostate specific antigen (PSA) level and Response Evaluation Criteria in Solid Tumors (RECIST) for measurable lesions, as assessed using Pearson's or Spearman's correlation coefficient. The relationship of changes in SUVmax and SULpeak with clinical response categories will also be assessed graphically and summarized overall with Spearman's rank correlation coefficient. Clinical response categories will be defined as complete response, partial response, stable disease, and progressive disease and determined by clinical assessment, conventional imaging, and biopsy (if available). The subgroup analysis of this group will be exploratory. Changes in uptake will be compared among all groups using ANOVA or the Kruskal-Wallis test and between pairs of groups using the t-test or Wilcoxon rank-sum test.
Change in 68Ga-PSMA-11 SULpeak | Baseline up to 6 weeks after systemic therapy initiation
  Expressed as percent (%) change from scan 1. Will be determined and correlated with change in prostate specific antigen (PSA) level and Response Evaluation Criteria in Solid Tumors (RECIST) for measurable lesions, as assessed using Pearson's or Spearman's correlation coefficient. The relationship of changes in SUVmax and SULpeak with clinical response categories will also be assessed graphically and summarized overall with Spearman's rank correlation coefficient. Clinical response categories will be defined as complete response, partial response, stable disease, and progressive disease and determined by clinical assessment, conventional imaging, and biopsy (if available). The subgroup analysis of this group will be exploratory. Changes in uptake will be compared among all groups using ANOVA or the Kruskal-Wallis test and between pairs of groups using the t-test or Wilcoxon rank-sum test.
Change in size of measurable metastatic lesions | Baseline up to 5 years post-scan
  Assessed by CT or magnetic resonance imaging (MRI) by RECIST 1.1 criteria.
Histopathologic demonstration of prostate cancer within biopsy or surgical resection specimens | Up to 5 years post-scan
  Will be performed only in patients with biopsy or surgical resection specimens. Lesions on each scan will be categorized as positive or negative. Pathology results will also be scored as positive or negative based on the clinical interpretation. These results will then be used to calculate accuracy with 95% CIs. CIs will be calculated using the non-parametric bootstrap with resampling by patient to account to dependence between lesions from the same patient.
Change in PSMA total tumor volume | Baseline up to 5 years post-scan
  Response defined by RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine L. Chen, M.D., Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No